CLINICAL TRIAL: NCT05387694
Title: Study of the Prognostic Value of the Coagulolytic Balance Dependent on Circulating Microvesicles in the Occurrence of Thrombotic Events After Total Knee Replacement in Orthopedic Surgery.
Acronym: MOTiVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A00582-41
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Knee Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Knee prosthesis group (Experimental)
  Interventions: Other: Thrombotic risk assessment

INTERVENTIONS:
Other: Thrombotic risk assessment — Collection of symptomatic thrombotic events occurring during the 5 days of hospitalization and then by telephone interview at M1 +/- 3 days. Complete echodoppler (proximal and distal) performed at M1 to highlight asymptomatic thrombotic events.

SUMMARY:
This is a prospective multicenter cohort study to evaluate the prognostic value of new biological markers in predicting thrombotic events after orthopedic surgery. According to the inclusion and non-inclusion criteria below, the study will include 387 major subjects who will undergo first-line total knee replacement and will receive the same standard prophylactic treatment: anticoagulation with Lovenox® (enoxaparin) 4000 IU/d subcutaneously 6 to 8 hours postoperatively and then daily for 15 days in combination with compression stockings.

DETAILED DESCRIPTION:
Recruitment and follow-up of patients will be carried out in 3 hospitals by the respective orthopedic teams. Three hundred and eighty-seven patients will be included in the study, over a period of 36 months: 200 in Marseille, 100 in Nice and 87 in Nîmes.

The objective of the study was to evaluate the prognostic capacities of the coagulolytic balance of MVs measured after surgery at D0 in the occurrence of a symptomatic or asymptomatic venous thromboembolic event revealed by echodoppler at 1 month after total knee replacement surgery.

The management of the subjects is unchanged from the current recommendations and will be homogeneous between the three inclusion centers. Patients will be hospitalized for 5 days and will receive the usual prophylactic anticoagulant treatment with Lovenox® (enoxaparin sodium; LMWH) 4000 IU/d subcutaneously 6 to 8 hours postoperatively and then daily for 15 days in combination with compression stockings, which corresponds to the management of a PTG according to current recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, aged 18 to 85 years (upper age limit classically used in the literature of PTG79-81)
* First-line TKP (knee native to any prosthesis) performed to treat primary or secondary osteoarthritis.

In case of contralateral PTG, a delay of 12 months between the 2 prostheses will be respected according to the habits of the inclusion centers.

* ASA score <4 (American Society of Anesthesiologists)
* No contraindication to prophylactic treatment with low molecular weight heparin (LMWH)
* Subject not taking anticoagulant or antiaggregant therapy at therapeutic dose
* Subject who has signed the informed consent form
* Subject affiliated to the social security system

Exclusion Criteria:

* Subjects with a history of sepsis, tumor or trauma in the considered joint
* Subject with sepsis or acute infection
* Immunocompromised subject (HIV, transplant, chemotherapy, leukemia, glucocorticoids >3 months)
* Subjects with severe respiratory, circulatory or cardiac pathologies involving anticoagulant treatment likely to influence the coagulolytic balance.
* Subject with severe renal insufficiency (creatinine clearance < 30ml/min)
* Subject refusing to participate in the study or not signing the informed consent or unable to adhere to the study procedures
* Subjects who are minors, pregnant or breastfeeding, not affiliated with the social security system, or deprived of liberty
* Subject already included in an interventional trial (which may alter the results of that study)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Area under the Receiver Operating Characteristic curve | After surgery at Day 0
  To assess the prognostic value of the microvesicle-dependent coagulolytic balance measured after D0 surgery (pre-administration of prophylactic treatment) in the occurrence of a post-total knee replacement thrombotic event (distal or proximal).

SECONDARY OUTCOMES:
Best prognostic threshold of MV coagulolytic balance measured | After surgery at Day 0
  Maximize sensitivity and specificity (Youden's method), and intrinsic and extrinsic performances associated with the threshold: sensitivity, specificity, positive likelihood ratio, negative likelihood ratio, positive predictive value, negative predictive value, with their 95% confidence intervals.
Estimation of the area under the ROC curve with its 95% confidence interval - The procoagulant activity of MV is dependent on FT | Day 0, Day 3 and 1 month post-PTG
  To assess the overall prognostic value of FT-dependent MV procoagulant activity at D0 (pre- and post-surgery) and D3, for the occurrence of a symptomatic or asymptomatic thrombotic event at 1 month post-PTG, the best prognostic threshold, and the intrinsic and extrinsic performance associated with the determined threshold, together with their 95% confidence intervals
Estimation of the area under the ROC curve with its 95% confidence interval - Fibrinolytic activity of MV | Day 0, Day 3 and 1 month post-PTG
  Allows assessment of the overall prognostic value of MV fibrinolytic activity at D0 (pre- and post-surgery) and D3, for the occurrence of a symptomatic or asymptomatic thrombotic event at 1 month post-PTG, best prognostic threshold, and intrinsic and extrinsic performance associated with the determined threshold, together with their 95% confidence interval.
Estimation of the area under the ROC curve with its 95% confidence interval - Coagulolytic balance of MV | Day 0, Day 3 and 1 month post-PTG
  Allows assessment of the prognostic value of the coagulolytic balance of MVs at D0 (before and after surgery) and D3, for the occurrence of a symptomatic thrombotic event (pulmonary embolism or DVT) at 1 month post-PTG, the best prognostic threshold, and the intrinsic and extrinsic performances associated with the determined threshold, together with their 95% confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique Hopitaux De Marseille; Matthieu OLLIVIER, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, Bouches Du Rhône, France